CLINICAL TRIAL: NCT07002216
Title: A Phase 2 Trial of Abbreviated Brentuximab Vedotin, Etoposide, Cyclophosphamide, Adriamycin, Dacarbazine, and Dexamethasone (BrECADD) Therapy in Stage 2 B-IV Hodgkin Lymphoma
Brief Title: BrECADD Therapy in Stage 2 B-IV Hodgkin Lymphoma
Acronym: BrECADD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Michele Stanchina, DO, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250293
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hodgkin Lymphoma; Advanced Hodgkin Lymphoma
Keywords: Stage 2 B-IV Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Etoposide; Cyclophosphamide; Doxorubicin; Dacarbazine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BrECADD (Brentuximab Vedotin, Etoposide, Cyclophosphamide, Doxorubicin, Dacarbazine, Dexamethasone) (Experimental): Participants in this group will receive each component of the BrECADD regimen at the recommended dosage listed in the United States Package Inserts (USPIs).
  Total participation duration is up to 24 months (2 years).
  Interventions: Drug: Brentuximab Vedotin; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Dacarbazine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Brentuximab Vedotin — Participants will receive 1.8 mg/kg of Brentuximab Vedotin intravenously (IV) for up to 30 minutes on Day 1 of each 21-day cycle period for up to 4 cycles in accordance with institutional procedures.
Drug: Etoposide — Participants will receive 150 mg/m^2 of Etoposide intravenously (IV) for up to 60 minutes on Days 1-3 of each 21-day cycle period for up to 4 cycles in accordance with institutional procedures.
Drug: Cyclophosphamide — Participants will receive 1250 mg/m^2 of Cyclophosphamide intravenously (IV) for up to 60 minutes on Day 1 of each 21-day cycle period for up to 4 cycles in accordance with institutional procedures.
Drug: Doxorubicin — Participants will receive 40 mg/m^2 of Doxorubicin intravenously (IV) for up to 30 minutes on Day 1 of each 21-day cycle period for up to 4 cycles in accordance with institutional procedures.
Drug: Dacarbazine — Participants will receive 250 mg/m^2 of Dacarbazine intravenously (IV) for up to 120 minutes on Days 2-3 of each 21-day cycle period for up to 4 cycles in accordance with institutional procedures.
Drug: Dexamethasone — Participants will self-administer 40 mg of Dexamethasone orally on Days 1-4 of each 21-day cycle period for up to 4 cycles in accordance with institutional procedures.

SUMMARY:
The purpose of this study is to further assess the efficacy and tolerability of a regimen of Brentuximab Vedotin, Etoposide, Cyclophosphamide, Doxorubicin, Dacarbazine, and Dexamethasone (BrECADD) in patients with Stage 2 B-IV Hodgkin Lymphoma (HL) with an exploratory objective to assess the clinical utility of Circulating tumor DNA (ctDNA) as a biomarker for minimal residual disease (MRD) and depth of treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years of age and ≤60 years of age on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place).
2. Patients must have histologic confirmation of classical Hodgkin Lymphoma (cHL) defined by the World Health Organization (WHO) classification.
3. Baseline Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) Computed Tomography (CT) must demonstrate Fluorodeoxyglucose (FDG) avid lesions compatible with computed tomography (CT)-defined anatomical tumor sites. Patients should have at least 1 measurable site of disease per Lugano classification in Fluorodeoxyglucose Positron Emission Tomography-Computed Tomography (FDG-PET/CT) or CT scans.
4. Patients must have a clinical stage consistent with:

   a. Stage 2 B cHL with one or both of the following risk factors: i. Large mediastinal mass (≥1/3 of the maximum transverse thoracic diameter) ii. Extranodal disease b. Stage III or Stage IV cHL based on Lugano criteria based on FDG-PET/CT.
5. Eastern Cooperative Oncology Group (ECOG) performance score (PS)≤ 2, except due to lymphoma involvement.
6. Life expectancy ≥3 months.
7. Women should avoid becoming pregnant for the full duration of chemotherapy and for up to 6 months after ending treatment. Therefore, women of childbearing potential must use highly effective contraceptive measures during treatment and for up to 6 months after stopping treatment. It is currently unknown whether brentuximab vedotin may reduce the effectiveness of hormonal contraceptives, and therefore, women using hormonal contraceptives should add a barrier method. Pregnancy testing is recommended for women of reproductive potential prior to initiating therapy.

   Agreement to use contraception during study participation.
   1. Female patients of childbearing potential must use highly effective methods of contraception.
   2. Patients using hormonal contraceptives (eg, birth control pills or devices) must use a barrier method of contraception (eg, condoms) as well.
   3. A woman is considered of childbearing potential, ie, fertile, following menarche and until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.
   4. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause.
8. Male patients with a female partner of childbearing potential are eligible if they abstain from sexual intercourse, are vasectomized, or if they agree to the use of barrier contraception with other methods described above during the study treatment period and for 120 days after the last dose of brentuximab vedotin.
9. Patients must have normal organ and marrow function as defined below:

   1. Absolute neutrophil count (ANC) >1,000 cells/mm3 independent of growth factor support within 7 days of study entry (≥750 cells/mm3 if lymphoma involvement of the bone marrow or spleen).
   2. Platelets ≥75,000 platelets/mm3 independent of transfusion support within 7 days of study entry (≥50,000 platelets/mm3 independent of transfusion support within 7 days of study entry if lymphoma involvement of the bone marrow or spleen).
   3. Hemoglobin >9 g/dL or >8 g/dL in case of bone marrow involvement by lymphoma independent of transfusion support within 7 days of study entry.
   4. Serum total bilirubin ≤2x upper limit of normal (ULN; except patients with Gilberts syndrome).
   5. Aspartate aminotransferase (AST; serum glutamic-oxaloacetic transaminase) and alanine transaminase (ALT; serum glutamic-pyruvic transaminase) ≤2.5x institutional ULN (≤3x institutional ULN if lymphoma involvement of the liver).
   6. Creatinine within normal institutional limits or creatinine clearance ≥40 mL/min (as estimated by the Cockcroft-Gault equation or alternative formula according to institutional guidelines) for patients with creatinine levels above institutional normal.
10. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments (SoA).

Exclusion Criteria:

1. Stage I or Stage IIA (IIA) HL.
2. Nodular lymphocyte-predominant HL.
3. Prior systemic lymphoma therapy including prior treatment with brentuximab vedotin.

   Note: Patients with prior treatment for indolent lymphoma are still eligible for participation as long as they did not receive anthracycline-based therapy.
4. Any uncontrolled or clinically significant cardiovascular disease including the following:

   1. Myocardial infarction within 6 months before screening;
   2. Unstable angina within 3 months before screening;
   3. New York Heart Association class III or IV congestive heart failure;
   4. History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes).
   5. Uncontrolled hypertension as indicated by ≥2 consecutive blood pressure measurements showing systolic blood pressure >170 mm Hg and/or diastolic blood pressure >105 mm Hg at screening.
5. Active and/or ongoing autoimmune anemia and/or autoimmune thrombocytopenia (eg, idiopathic thrombocytopenia purpura).
6. Uncontrolled concurrent illness, such as liver cirrhosis, diabetes, autoimmune disorder requiring immunosuppression or long-term corticosteroids (>10 mg daily prednisone equivalent), or any other serious medical condition, laboratory abnormality, or psychiatric illness which would compromise ability to comply with study procedures.
7. Severe or debilitating pulmonary disease.
8. Peripheral neuropathy ≥Grade 2.
9. Concurrent malignancy requiring active therapy.
10. Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancer.
11. Active fungal, bacterial and/or viral infection requiring systemic therapy.
12. Breastfeeding or pregnant women.
13. Known active infection with human immunodeficiency virus (HIV), or serologic status reflecting active hepatitis B or C infection as follows:

    1. Patients with positive HIV test and undetectable viral load will be eligible for this study.
    2. Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb): Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (<20 IU), and if they are willing to undergo monitoring every 4 weeks for HBV reactivation.
    3. Presence of hepatitis C virus (HCV) antibody: Patients with presence of HCV antibody are eligible if HCV ribonucleic acid (RNA) is undetectable.
14. Patients with impaired decision-making capacity.
15. Underlying medical conditions that, in the Investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs.
16. Patients undergoing major surgery ≤4 weeks prior to receiving their first dose of BrECADD. Major surgery is defined as open-heart, reconstructive, transplant, removal of a brain tumor, or a damaged kidney surgery.
17. Vaccination or requirement for vaccination with a live vaccine within 28 days prior to the first dose of study drug or at any time during planned study treatment.
18. Hypersensitivity to brentuximab vedotin, any components of the BrECADD regimen, or any of the other ingredients of the applicable study medications.
19. Concurrent participation in another therapeutic clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2030-07-15 (Estimated); Study Completion 2030-07-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 12 months
  Progression-free survival (PFS) is defined as the elapsed time in months from the start of treatment until disease progression or death, whichever is earlier. Follow-up times for participants who remain alive without progression will be censored at the last documented disease assessment date.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  Progression-free survival (PFS) is defined as the elapsed time in months from the start of treatment until disease progression or death, whichever is earlier. Follow-up times for participants who remain alive without progression will be censored at the last documented disease assessment date.
Number of Treatment-Related Adverse Events (AEs) | Up to 40 months
  The number of treatment-related AEs will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0. Standard definitions for seriousness will be applied.
Number of Treatment-Related Serious Adverse Events (SAEs) | Up to 40 months
  The number of treatment-related SAEs will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0. Standard definitions for seriousness will be applied.
Percentage of Participants With Toxicity Throughout BrECADD Measured by PRO-CTCAE | Up to 40 months
  Toxicity will be measured by the percentage of participants using the Participant Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE). This criteria is a measurement system designed by the National Cancer Institute (NCI) to capture and evaluate the symptomatic side effects experienced by cancer patients during clinical trials, allowing patients to self-report on the frequency, severity, interference, and presence/absence of symptoms like pain, fatigue, nausea, and skin reactions, providing a more patient-centric perspective on treatment toxicity compared to clinician-based assessments alone.
Percentage of Participants With Toxicity Throughout BrECADD measured by FRAIL | Up to 40 months
  Toxicity will be measured by the percentage of participants using the Fatigue, Resistance, Aerobic Capacity, Illnesses and Loss of Weight (FRAIL) questionnaire.
  The FRAIL scale (short five-questions assessment of fatigue, resistance, aerobic capacity, illnesses and loss of weight) classified the patients into three categories: robust (score=0), pre-frailty (score=1-2), and frailty (score=3-5)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Stanchina, DO, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No